CLINICAL TRIAL: NCT03155308
Title: Validation of the NICE Classification Using Pentax Chromoendoscopy (I-scan and Optical Enhancement System
Brief Title: Validation of the NICE Classification Using Pentax Chromoendoscopy
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: MAY 2-2017
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — colorectal polyps will be resected y biopsed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polyp group: Consecutive adult patients between 18 and 80 years of age, referred for elective outpatient colonoscopy and in whom polypectomy or biopsy is perform will be enrolled to be evaluated using Pentax chromoendoscopy (i-scan and Optical Enhancement)
  Interventions: Device: Pentax chromoendoscopy (i-scan and Optical Enhancement)

INTERVENTIONS:
Device: Pentax chromoendoscopy (i-scan and Optical Enhancement) — All lesions will be evaluated using the 3 i-scan modes and the 2 OE modes without magnification. The lesion size data, location and macroscopic shape of the lesions based on the Paris classification will be recorded. Finally all lesions will be classified in real-time into 3 types based on NICE classification (NICE 1, hyperplastic polyps; NICE 2, adenoma and superficial submucosal carcinoma; NICE 3, SM-d invasive carcinoma). A level of confidence (high or low) will be assign in each stage. Polyp's images will be photographically and videotape recorded. All polyps will be resected or biopsied for histopathological examination used as the criterion standard for the analysis.

SUMMARY:
Colorectal cancer (CRC) is the most frequent gastrointestinal tumor and the second cause of cancer related death. Colonoscopy is currently the recommended method for detection of polyps and cancers in the colon. Removal of all adenomatous polyps during colonoscopy has become worldwide a standard procedure as it has been demonstrated to significantly reduce colorectal cancer incidence and mortality. It is routine practice to remove all the detected polyps for pathological evaluation, due to the low accuracy (59% to 84%) to differentiate non-neoplastic from neoplastic colorectal lesions with white-light endoscopy. The development of electronic or virtual chromoendoscopy (CE) has aimed to reliably predict histology of colorectal lesions based on endoscopic features. This technology differentiates between neoplastic and non-neoplastic lesions base on the analysis of the neo-angiogenesis and the mucosal pit pattern. Optical endoscopic diagnosis allows the real-time evaluation of polyp histology during colonoscopy and to determine the appropriate therapeutic strategy. This is important in clinical practice, since adenomas or superficial invasive submucosal carcinoma lesions can be curatively treated by endoscopic removal, unlike deeply invasive carcinomas, which requires surgery. The Narrow-band imaging (NBI) international colorectal endoscopic (NICE) classification is validated classification system proposed as a valid tool for not only differentiating hyperplastic from adenomatous polyps, but also predicting submucosal deep (SM-d) carcinomas. It was developed based on NBI technology, leaving uncertainty on its applicability to other systems. It was previously evaluated the application of the NICE classification to Fujinon spectral Imaging Color Enhancement (FICE) technology founding suboptimal results (accuracy 77%, sensitivity 77% and specificity 75%) and moderate inter-observer agreement (kappa: 0.51).

DETAILED DESCRIPTION:
NBI technology uses a physical filter in order to exploit the capacity of hemoglobin to selectively absorb blue light. It is considered to be less useful in areas with a large lumen, such as the stomach and colon, as a result of insufficient light for wide-range observation of the full extent of the tissue surface, and because the images are dark. I-scan is a virtual chromoendoscopy, based on the principle of digital post-processing and consists of three different image algorithms. Mode 1 is for detection of lesions. This algorithm is used for surface enhancement (SE) and enhances light-dark contrast by obtaining luminance intensity data for each pixel and apply an algorithm that allows detailed observation of the mucosal surface structure and lesion borders without altering the brightness of the endoscopic picture. Mode 2 is for characterization of lesions. This algorithm combines SE and tone enhancement (TE). TE dissects and analyses the individual red-green-blue components of a normal endoscopic image in real time and then alters the color frequencies of each component and recombines the components to a single, new color image without visible delay for the examiner. It is used to enhance minute mucosal changes and vessel structures. Mode 3 adds contrast enhancement (CE) to the endoscopic image (in addition to SE and TE) and is for demarcation of lesions. It digitally adds blue color to dark areas within the endoscopic image. Recently an image-enhanced endoscopic technology using a pre-processor band-limited light called Optical Enhancement system (OE system™), was developed by HOYA Co. (Tokyo, Japan) and is now equipped with the latest endoscopy system (Pentax Video Processor EPK-i7010; HOYA Co.). This new technology combines digital signal processing with optical filters that overcomes the limit of the spectral characteristics of the illumination light. Previous i-scan technology uses white light alone as an illumination light and digital post-processing of the reflection afterwards creates images yielding the virtual chromoendoscopic image. Although accumulating evidence has shown the usefulness of i-scan in the clinical setting, emission of white light alone causes a potential limitation for the current i-scan technology to obtain higher contrast images of microvascular pattern on the mucosal surface as shown by Narrow Band Imaging (NBI). The basic concept of OE is to overcome the darkness of NBI, which results in less usefulness for detectability in wide-range observation in the full-extended gastrointestinal lumen. The new innovated optical filters achieve higher illumination intensity and overall transmittance by connecting the peaks of the hemoglobin absorption spectrum (415 nm, 540 nm and 570 nm) creating a continuous wavelength spectrum. There are two modes with different OE filters. Mode 1 is designed mainly to improve visualization of microvessels with a sufficient amount of light, and Mode 2 is designed to improve contrast of white-light observation by bringing the color tone of the overall image closer to that of natural color (white color tone). Due to the underlying differences between the NBI and Pentax technologies (i-scan and OE system), it remains uncertain whether the NICE classification may be translated to this technology. The aim of this study is to validate the NICE classification by applying i-scan and OE system with high-definition without optical magnification, to evaluate colorectal lesions.

MATERIALS AND METHODS

Study design: It will be a non-interventional, prospective, non-randomized, non-controlled and simple blind study, performed in the Ecuadorian Institute of Digestive Disease (IECED), OmniHospital Academic Tertiary Center Ecuador, with patients included from April 2017 to October 2017. The study protocol and consent form has been approved by the institutional review board and will be conducted according to the declaration of Helsinki. Written informed consent will be obtained from all subjects before the examination.

Study Population: Consecutive adult patients between 18 and 80 years of age, referred for elective outpatient colonoscopy and in whom polypectomy or biopsy is performed will be enrolled. Exclusion criteria will be pregnancy, suspected colonic obstruction or history of previous obstruction, gastrointestinal bleeding, history colorectal surgery, inflammatory bowel disease, hereditary polyposis syndrome, diverticulitis, history of radiation therapy to abdomen or pelvis, history of severe cardiovascular, pulmonary, liver or renal disease, severe coagulation disorders or use of anticoagulants. Patients with polyps but in whom histopathology has not been evaluated or with a poor bowel preparation (Boston Bowel Preparation Scale ≤6) will be excluded from the analysis but included in the intention to treat.

Intervention: endoscopic technique The procedures will be performed under propofol intravenous sedation, in left later or supine position. For bowel preparation, the participants will have to ingest 4 liters of polyethylene glycol solution in the evening the day before the procedure. The effectiveness of the bowel cleansing will be evaluated using the Boston Bowel Preparation Scale. Three colonoscopists (C.R.M., M.V., M.S.A.), with extensive experience in colonoscopy with i-scan and OE (>1000 cases) and familiar with the NICE classification, will perform the procedures using Pentax high definition colonoscopes without optical magnification (EC-3890Zi, PENTAX Medical, HOYA Co.) and EPK-i7010 processor with the ability to display i-scan and OE system™ images. The endoscopy images will be analyzed on a 27-inch, flat panel, high definition LCD monitors (Radiance™ ultra SC-WU27-G1520 model). All lesions initially detected by white light endoscopy will be intensively washed using a water ejection pump before recording the procedure and then the endoscopic features on the surface will be evaluated using the 3 i-scan modes and the 2 OE modes without magnification. The lesion size data (1-5/6-9/>10 mm), location (cecum/ right/ transverse/ left/ sigmoid colon/ rectum) and macroscopic shape of the lesions based on the Paris classification will be recorded. The size will be estimated with biopsy forceps (2.2 mm closed; Radial Jaw 4, Boston Scientific, Marlborough, Massachusetts, USA) or polypectomy snare (13mm open; Captivator, Boston Scientific, Marlborough, Massachusetts, USA). Finally all lesions will be classified in real-time into 3 types based on NICE classification (NICE 1, hyperplastic polyps; NICE 2, adenoma and superficial submucosal carcinoma; NICE 3, SM-d invasive carcinoma). A level of confidence (high or low) will be assign in each stage. A high confidence prediction will be considered when the endoscopist is 90% certain of the diagnosis and this condition will be consider when polyps have ≥1 features associated with one NICE type and no features associated to the others NICE type. If there are uncertainty regarding the features or if there are features from different NICE types the prediction will have low confidence. Polyp's images will be photographically and videotape recorded. Each high-definition video will consist of 30 to 60 seconds of white-light endoscopy followed by i-scan 1,2,3 and OE mode 1 and 2. For the purpose of this study, magnification was not allowed during recording. All polyps will be resected or biopsied for histopathological examination used as the criterion standard for the analysis. Two experienced pathologists, blind to the endoscopic diagnosis, will assess the histology according to the revised Vienna classification. Lesions identified histopathologically as serrated adenomas/ polyps or traditional serrated adenoma will be excluded from the analysis but included in the intention to treat, due to the lack of fully established evidence of NICE classification utility for the diagnosis of these lesions.

In a second phase, endoscopists with less experience (<1000 procedures) using i-scan and OE will be selected. After a formal instruction on the NICE classification based on theoretical background and a series of i-scan/OE-polyp images, each of them will have to reviewed all the videos and applied the NICE classification in order to predict the histology. Each of the three criteria of the NICE system (colour/vessel/surface pattern) will be individually scored as well as the overall level of confidence (high/low).

Statistical analysis

Base line characteristics will be expressed as percentage or mean +/- standard deviation. It will be calculated the accuracy, sensitivity, specificity, negative and positive predictive values with the 95% of Confidence Interval (95% CI), for each component of the classification and for the overall prediction by using the classification. Using multilevel logistic regression, the sensitivity and specificity of the different criteria, will be compared. Diagnostic values of the criteria used in combination (combination of "at least 1 criterion being positive" versus "all combined criteria being positive") will be assessed and compared. The criterion standard for validation of predictions will be the lesions histology. Presence of adenomatous feature at each criterion will be defined as a positive result. The sample size was calculated assuming that 80% of predictions will be made with high confidence, and that the real accuracy will be 90%. A data set containing 30 random-selected videos will be presented after 2 months to the three main investigators (C.R.M, M.V, M.S.A.) in order to assess intra and inter-observer reproducibility. The endoscopists will have classified again the polyps according to the three types on the NICE classification. To examine inter and intra observer agreement, kappa values will be calculated. Kappa coefficients below 0.4 indicate "poor agreement," values between 0.4 and 0.8 represent "moderate to good agreement," and values greater than 0.8 indicate "excellent agreement." A P value of less than 0.05 will be considered to be statistically significant. All the statistical analysis will be performed using SPSS software suite v.22.

ELIGIBILITY:
Inclusion Criteria: Consecutive adult patients between 18 and 80 years of age, referred for elective outpatient colonoscopy and in whom polypectomy or biopsy is performed will be enrolled.

Exclusion Criteria: pregnancy, suspected colonic obstruction or history of previous obstruction, gastrointestinal bleeding, history colorectal surgery, inflammatory bowel disease, hereditary polyposis syndrome, diverticulitis, history of radiation therapy to abdomen or pelvis, history of severe cardiovascular, pulmonary, liver or renal disease, severe coagulation disorders or use of anticoagulants.

Patients with polyps but in whom histopathology has not been evaluated or with a poor bowel preparation (Boston Bowel Preparation Scale ≤6) will be excluded from the analysis but included in the intention to treat.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients between 18 and 80 years of age, referred for elective outpatient colonoscopy and in whom polypectomy or biopsy is performed will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Pentax chromoendoscopy (i-scan and Optical Enhancement system) for differentiating between the three types of NICE classification. | 4 month
  colorectal polypoid lesions will be evaluated using Pentax chromoendoscopy (i-scan and OE system) in order to classified the lesions by NICE classification. The histopathology will be evaluated from all lesions as Gold Standard and finally accuracy, sensitivity, specificity, positive predictive value and negative predictive value will be calculated.

SECONDARY OUTCOMES:
assessment of inter- and intra-observer agreement | 4 month
  A data set containing 30 random-selected videos will be presented after 2 months to the three main investigators (C.R.M, M.V, M.S.A.) in order to assess intra and inter-observer reproducibility. The endoscopists will have classified again the polyps according to the three types on the NICE classification. To examine inter and intra observer agreement, kappa values will be calculated. Kappa coefficients below 0.4 indicate "poor agreement," values between 0.4 and 0.8 represent "moderate to good agreement," and values greater than 0.8 indicate "excellent agreement."
Diagnostic accuracy of the individual criteria of NICE classification using i-scan and OE system. | 4 month
  It will be calculated the accuracy, sensitivity, specificity, negative and positive predictive values with the 95% of Confidence Interval (95% CI), for each component of the classification and for the overall prediction by using the classification. Using multilevel logistic regression, the sensitivity and specificity of the different criteria, will be compared. Diagnostic values of the criteria used in combination (combination of "at least 1 criterion being positive" versus "all combined criteria being positive") will be assessed and compared. The criterion standard for validation of predictions will be the lesions histology. Presence of adenomatous feature at each criterion will be defined as a positive result.
Diagnostic accuracy according to the level of confidence. | 4 month
  A level of confidence (high or low) will be assign in each stage. A high confidence prediction will be considered when the endoscopist is 90% certain of the diagnosis and this condition will be consider when polyps have ≥1 features associated with one NICE type and no features associated to the others NICE type. If there are uncertainty regarding the features or if there are features from different NICE types the prediction will have low confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Madranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Cancer Statistics Working Group. United States Cancer Statistics: 1999 - 2005 Incidence and Mortality Web-Based Report. US Department of Health and Human Services, Centers for Disease Control and Prevention and National Cancer Institute: Atlanta, 2009
- [Background] Gono K, Yamazaki K, Doguchi N et al. Endoscopic observation of tissue by narrow band illumination. Opt. Rev. 2003; 10: 211-5.
- [Result] Rex DK, Johnson DA, Anderson JC, Schoenfeld PS, Burke CA, Inadomi JM; American College of Gastroenterology. American College of Gastroenterology guidelines for colorectal cancer screening 2009 [corrected]. Am J Gastroenterol. 2009 Mar;104(3):739-50. doi: 10.1038/ajg.2009.104. Epub 2009 Feb 24. PMID 19240699
- [Result] Levin B, Lieberman DA, McFarland B, Andrews KS, Brooks D, Bond J, Dash C, Giardiello FM, Glick S, Johnson D, Johnson CD, Levin TR, Pickhardt PJ, Rex DK, Smith RA, Thorson A, Winawer SJ; American Cancer Society Colorectal Cancer Advisory Group; US Multi-Society Task Force; American College of Radiology Colon Cancer Committee. Screening and surveillance for the early detection of colorectal cancer and adenomatous polyps, 2008: a joint guideline from the American Cancer Society, the US Multi-Society Task Force on Colorectal Cancer, and the American College of Radiology. Gastroenterology. 2008 May;134(5):1570-95. doi: 10.1053/j.gastro.2008.02.002. Epub 2008 Feb 8. PMID 18384785
- [Result] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Result] De Palma GD, Rega M, Masone S, Persico M, Siciliano S, Addeo P, Persico G. Conventional colonoscopy and magnified chromoendoscopy for the endoscopic histological prediction of diminutive colorectal polyps: a single operator study. World J Gastroenterol. 2006 Apr 21;12(15):2402-5. doi: 10.3748/wjg.v12.i15.2402. PMID 16688833
- [Result] Fu KI, Sano Y, Kato S, Fujii T, Nagashima F, Yoshino T, Okuno T, Yoshida S, Fujimori T. Chromoendoscopy using indigo carmine dye spraying with magnifying observation is the most reliable method for differential diagnosis between non-neoplastic and neoplastic colorectal lesions: a prospective study. Endoscopy. 2004 Dec;36(12):1089-93. doi: 10.1055/s-2004-826039. PMID 15578300
- [Result] Su MY, Hsu CM, Ho YP, Chen PC, Lin CJ, Chiu CT. Comparative study of conventional colonoscopy, chromoendoscopy, and narrow-band imaging systems in differential diagnosis of neoplastic and nonneoplastic colonic polyps. Am J Gastroenterol. 2006 Dec;101(12):2711-6. doi: 10.1111/j.1572-0241.2006.00932.x. PMID 17227517
- [Result] Kudo S, Tamura S, Nakajima T, Yamano H, Kusaka H, Watanabe H. Diagnosis of colorectal tumorous lesions by magnifying endoscopy. Gastrointest Endosc. 1996 Jul;44(1):8-14. doi: 10.1016/s0016-5107(96)70222-5. PMID 8836710
- [Result] Kato S, Fujii T, Koba I, Sano Y, Fu KI, Parra-Blanco A, Tajiri H, Yoshida S, Rembacken B. Assessment of colorectal lesions using magnifying colonoscopy and mucosal dye spraying: can significant lesions be distinguished? Endoscopy. 2001 Apr;33(4):306-10. doi: 10.1055/s-2001-13700. PMID 11315890
- [Result] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Result] Machida H, Sano Y, Hamamoto Y, Muto M, Kozu T, Tajiri H, Yoshida S. Narrow-band imaging in the diagnosis of colorectal mucosal lesions: a pilot study. Endoscopy. 2004 Dec;36(12):1094-8. doi: 10.1055/s-2004-826040. PMID 15578301
- [Result] Apel D, Jakobs R, Schilling D, Weickert U, Teichmann J, Bohrer MH, Riemann JF. Accuracy of high-resolution chromoendoscopy in prediction of histologic findings in diminutive lesions of the rectosigmoid. Gastrointest Endosc. 2006 May;63(6):824-8. doi: 10.1016/j.gie.2005.09.013. PMID 16650546
- [Result] Tischendorf JJ, Wasmuth HE, Koch A, Hecker H, Trautwein C, Winograd R. Value of magnifying chromoendoscopy and narrow band imaging (NBI) in classifying colorectal polyps: a prospective controlled study. Endoscopy. 2007 Dec;39(12):1092-6. doi: 10.1055/s-2007-966781. PMID 18072061
- [Result] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Result] Hayashi N, Tanaka S, Hewett DG, Kaltenbach TR, Sano Y, Ponchon T, Saunders BP, Rex DK, Soetikno RM. Endoscopic prediction of deep submucosal invasive carcinoma: validation of the narrow-band imaging international colorectal endoscopic (NICE) classification. Gastrointest Endosc. 2013 Oct;78(4):625-32. doi: 10.1016/j.gie.2013.04.185. Epub 2013 Jul 30. PMID 23910062
- [Result] Repici A, Ciscato C, Correale L, Bisschops R, Bhandari P, Dekker E, Pech O, Radaelli F, Hassan C. Narrow-band Imaging International Colorectal Endoscopic Classification to predict polyp histology: REDEFINE study (with videos). Gastrointest Endosc. 2016 Sep;84(3):479-486.e3. doi: 10.1016/j.gie.2016.02.020. Epub 2016 Feb 27. PMID 26928372
- [Result] Gono K, Obi T, Yamaguchi M, Ohyama N, Machida H, Sano Y, Yoshida S, Hamamoto Y, Endo T. Appearance of enhanced tissue features in narrow-band endoscopic imaging. J Biomed Opt. 2004 May-Jun;9(3):568-77. doi: 10.1117/1.1695563. PMID 15189095
- [Result] Kodashima S, Fujishiro M, Ono S, Niimi K, Mochizuki S, Asada-Hirayama I, Konno-Shimizu M, Matsuda R, Minatsuki C, Nakayama C, Takahashi Y, Sakaguchi Y, Yamamichi N, Tanaka C, Koike K. Evaluation of a new image-enhanced endoscopic technology using band-limited light for detection of esophageal squamous cell carcinoma. Dig Endosc. 2014 Mar;26(2):164-71. doi: 10.1111/den.12108. Epub 2013 Apr 29. PMID 23621480
- [Result] Neumann H, Fujishiro M, Wilcox CM, Monkemuller K. Present and future perspectives of virtual chromoendoscopy with i-scan and optical enhancement technology. Dig Endosc. 2014 Jan;26 Suppl 1:43-51. doi: 10.1111/den.12190. Epub 2013 Oct 23. PMID 24373000
- [Result] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Result] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Result] Quirke P, Risio M, Lambert R, von Karsa L, Vieth M. Quality assurance in pathology in colorectal cancer screening and diagnosis-European recommendations. Virchows Arch. 2011 Jan;458(1):1-19. doi: 10.1007/s00428-010-0977-6. PMID 21061133
- [Result] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Result] Kodashima S, Fujishiro M. Novel image-enhanced endoscopy with i-scan technology. World J Gastroenterol. 2010 Mar 7;16(9):1043-9. doi: 10.3748/wjg.v16.i9.1043. PMID 20205272